CLINICAL TRIAL: NCT00479505
Title: A Multi-Center, Randomised, Parallel Group, Double-Blind, Placebo Controlled Estimation Study To Assess The Efficacy And Safety Of Modified Release UK-369,003 In The Treatment Of Men With Storage Lower Urinary Tract Symptoms (LUTS) With And Without Erectile Dysfunction (ED).
Brief Title: Study The Effects Of Different Doses Of UK-369,003 In Men With Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3711047
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — 1-(6-ethoxy-5-(3-ethyl-6,7-dihydro-2-(2-methoxyethyl)-7-oxo-2H-pyrazolo(4,3-d)pyrimidin-5-yl)-3-pyridyl sulphonyl)-4-ethylpiperazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: UK-369,003
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UK-369,003 — UK-369,003 100mg, 50mg, 25mg and 10mg doses in addition to placebo.
  Arms: Active
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a 12 week study in which different doses of UK-369,003 will be administered to patients with a diagnosis of overactive bladder. Patients will complete a series of questionnaires before treatment, during treatment and after treatment, to assess whether UK-369,003 has improved their symptoms of overactive bladder and erectile function.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18 years and above
* documented clinical diagnosis of overactive bladder with urinary frequency >= 8 times / 24 hours and number of urgency episodes > 1 episode / 24 hours.

Exclusion Criteria:

* Neurological diseases known to affect bladder function.
* Urinary tract infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
This is an estimation study with no primary endpoint. There are efficacy endpoints. | 12 Weeks

SECONDARY OUTCOMES:
Patient reported treatment impact questionnaire. | 12 Weeks
Lower urinary tract symptoms diary. | 12 Weeks
International prostate symptom score questionnaire. | 12 Weeks
OAB-q short form questionnaire. | 12 Weeks
Patient perception of bladder control questionnaire. | 12 Weeks
International index of erectile function questionnaire. | 12 Weeks
International consultation on incontinence questionnaire. | 12 Weeks
Quality of erection questionnaire. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (49):
- Australia (2):
  - Pfizer Investigational Site, Miranda, New South Wales
  - Pfizer Investigational Site, Kippa-Ring, Queensland
- Canada (4):
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
- Chile (2):
  - Pfizer Investigational Site, Rancagua, Región del Libertador General Bernardo O’Higgins
  - Pfizer Investigational Site, Santiago, RM
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogota, Cundinamarca
- Finland (5):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kouvola
  - Pfizer Investigational Site, Oulu
  - Pfizer Investigational Site, Tampere
  - Pfizer Investigational Site, Turku
- France (5):
  - Pfizer Investigational Site, Garches
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rennes
- Germany (5):
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, Muelheim A.d. Ruhr
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Rosenheim
- Greece (3):
  - Pfizer Investigational Site, Cholargós, Athens
  - Pfizer Investigational Site, Epirus, Ioannina
  - Pfizer Investigational Site, Rio, Patras
- Italy (3):
  - Pfizer Investigational Site, Cefalù, Palermo
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Latina
- Pfizer Investigational Site, Riga, Latvia
- Norway (2):
  - Pfizer Investigational Site, Moelv
  - Pfizer Investigational Site, Oslo
- Poland (4):
  - Pfizer Investigational Site, Mysłowice
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Szczecin
  - Pfizer Investigational Site, Wroclaw
- Slovakia (4):
  - Pfizer Investigational Site, Bratislava, Slovakia
  - Pfizer Investigational Site, Martin, Slovakia
  - Pfizer Investigational Site, Trenčín, Slovakia
  - Pfizer Investigational Site, Košice
- Spain (2):
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Manacor, Palma de Mallorca
- Switzerland (2):
  - Pfizer Investigational Site, Aarau
  - Pfizer Investigational Site, Zurich
- United Kingdom (3):
  - Pfizer Investigational Site, High Heaton, Newcastle upon Tyne
  - Pfizer Investigational Site, Taunton, Somerset
  - Pfizer Investigational Site, Leeds

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3711047&StudyName=Study%20The%20Effects%20Of%20Different%20Doses%20Of%20UK-369%2C003%20In%20Men%20With%20Overactive%20Bladder.